CLINICAL TRIAL: NCT02744365
Title: Biobank of Data and of Human Biological Samples on Prematurity, Preeclampsia and Other Pregnancy Complications
Brief Title: Biobank on Prematurity, Preeclampsia and Other Pregnancy Complications
Status: Recruiting | Type: Observational
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Principal Investigator, Emmanuel Bujold, Professor, CHU de Quebec-Universite Laval
Other Study IDs: 2015-2272
Record Dates: First submitted 2016-04-15; First posted 2016-04-20 (Estimated); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Preeclampsia; Preterm Birth; Pregnancy Complications; Fetal Anomalies
MeSH Terms: conditions — Pre-Eclampsia; Premature Birth; Pregnancy Complications; Congenital Abnormalities | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — maternal plasma, maternal serum and buffy coat, maternal urine, cord blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Prediction Group: The women recruited in the biobank through the Prediction Study (NCT02189148) are low-risk pregnant women between 11 and 13 6/7 weeks of gestation (N=7600 maximum).
  Interventions: Other: Observational
- PEARL Group: The women recruited in the biobank through the PEARL Study (NCT02379832) are :
  1. low-risk pregnant women between 11 and 13 6/7 weeks of gestation (controls, N=45)
  2. pregnant women with diagnosis of preeclampsia between 20 and 41 6/7 weeks of gestation (cases, N=45)
  Interventions: Other: Observational
- GAP Group: The women recruited in the biobank through the GAP Trial (NCT02280031) are women pregnant with twins between 11 3/7 and 13 6/7 weeks of gestation(N=50 maximum) randomized for placebo or aspirin.
  Interventions: Other: Observational
- PREDICTION 2 Group: The women recruited in the biobank through the Prediction-2 Study (NCT03067298) are nulliparous pregnant women between 14 and 15 6/7 weeks of gestation (N=1000 maximum).
  Interventions: Other: Observational
- HAUPE Study: Women that are at risk of pre-eclampsia and great obstetrical syndroms (elevated maternal age, invitro fertilization, chronic disease) (N=60) and a control group not at risk (N=60)
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — All women of the biobank have provided:
  1. blood samples (plasma, serum and Buffy-coat)
  2. urine samples
  3. demographic and clinical data (maternal age, BMI, smoking status, obstetrical and medical history)
  4. mean arterial blood pressure
  5. ultrasound examination (datation of pregnancy at recruitment, uterine arteries doppler, placental volume, nuchal translucency in the majority of the cases)
  6. access to medical record (for pregnancy/delivery outcomes, newborn birthweight, gestational age at delivery)

SUMMARY:
The Biobank includes data and biological specimens of women from three original studies: 1) First-trimester Prediction of Preeclampsia (PREDICTION Study, NCT02189148), 2) Pre-Eclampsia And growth Retardation, an evaluative Longitudinal study (PEARL Study, NCT02379832), 3) Effect of Low Dose Aspirin on Birthweight in Twins: The GAP Trial (NCT02280031) and 4)PREDICTION2: Prediction of Preeclampsia and other Pregnancy Complications Following Combined Iterative Screening.

DETAILED DESCRIPTION:
This Biobank is comprised of: 1) medical, social, obstetrical and ultrasonographic data, 2) human biological samples (maternal plasma, serum and buffy coat, maternal urine, cord blood) and 3) the results derived from these (biochemical or ultrasonographic markers, genetics, risk calculations ...)

ELIGIBILITY:
Inclusion Criteria:

* (specific to each study)

Exclusion Criteria:

* pregnant women <18 years old at recruitment
* negative fetal heart at recruitment
* women not able to provide an informed consent to the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: According to each study:
  1. Prediction study: Nulliparous women between 11 and 13 6/7 weeks of gestation
  2. PEARL study: Nulliparous women between 11 and 13 6/7 weeks of gestation or diagnosed with preeclampsia between 20 and 42 weeks of gestation
  3. GAP Study: women with twin pregnancy between 11 and 13 6/7 weeks of gestation
  4. Prediction-2 study: Nulliparous women with singleton pregnancy without fetal anomaly/demise between 14 and 15 6/7 weeks of gestation
Sampling Method: Non-Probability Sample
Enrollment: 7845 (Estimated)
Dates: Start 2015-04 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
early onset preeclampsia | diagnosed between 20 and 34 weeks of gestation
  Preeclampsia will be defined according to the Canadian Guidelines for Diagnosis, Evaluation, and Management of the Hypertensive Disorders of Pregnancy guidelines, as de novo hypertension with diastolic blood pressure >90 mmHg on two occasions at least four hours apart, after 20 weeks of pregnancy, associated with proteinuria ≥300 mg/24 h or at least '2 +' protein on urine dipstick or an adverse conditions

SECONDARY OUTCOMES:
Severe preeclampsia | between 20 and 42 weeks of gestation
  Severe Preeclampsia will be defined by the presence of at least one of the following adverse condition: 1) systolic blood pressure ≥ 160 mmHg and diastolic blood pressure ≥ 110 mmHg after 4 h of bed rest, 2) proteinuria ≥ 5 g/24 h or at least '3 +' protein on urine dipstick, or 3) oliguria < 400 ml/24 h; 4) cerebral or visual disturbances; epigastric pain; pulmonary edema or cyanosis; thrombocytopenia <100,000mm
Fetal growth restriction | between 20 and 42 weeks of gestation
  Fetal growth restriction will be defined as a birth weight below the 10th centile (or below the 3rd centile for severe FGR) of Canadian reference growth charts.
spontaneous preterm birth | between 20 and 36 6/7 weeks of gestation
  sPTB is a birth occuring spontaneously between 20 and 36 6/7 weeks of gestation
Fetal aneuploidies | diagnosed during or after pregnancy
  Any fetal chromosome that has an abnormal number of copies. Example: trisomy 13, 18 or 21.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Bujold, MD, MSc, Principal Investigator — CHU de Quebec
Locations (1):
- CHU de Quebec, Québec, Canada

IPD SHARING:
Plan to Share IPD: Yes
We will publish the results linked to the data collected. We will share these data with other groups that are interested in research on preeclampsia and other pregnancy complications.